CLINICAL TRIAL: NCT00006121
Title: Phase II Study of Oxaliplatin Single Agent in Patients With Metastatic Breast Cancer After Failure of Anthracycline/Taxane Based Chemotherapy
Brief Title: Oxaliplatin in Treating Women With Advanced or Metastatic Breast Cancer That Has Not Responded to Previous Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16001-10005; EORTC-16001
Record Dates: First submitted 2000-08-03; First posted 2003-10-08 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage III breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating women who have advanced or metastatic breast cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of oxaliplatin in patients with advanced or metastatic breast cancer following failure of anthracycline/taxane based chemotherapy.
* Determine objective response, duration of response, and time to progression in these patients when treated with this regimen.
* Determine the acute side effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks until disease progression and then every 3 months for survival.

PROJECTED ACCRUAL: A total of 27-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or metastatic breast cancer
* Bidimensionally measurable disease

  * At least one lesion at least 2 cm in one dimension by CT scan or MRI
* Must have failed prior anthracycline/taxane based chemotherapy as defined by one of the following:

  * Stage IV disease treated with anthracycline/taxane combination as first line therapy for advanced or metastatic disease
  * Stage IV disease treated with first line anthracycline therapy and second line taxane therapy for advanced or metastatic disease
  * Any adjuvant treatment other than anthracycline based therapy followed by anthracycline/taxane combination as first line therapy for advanced or metastatic disease
  * Any adjuvant therapy other than anthracycline based therapy followed by first line anthracycline based therapy and second line taxane based therapy for advanced or metastatic disease
  * Adjuvant anthracycline based therapy followed by relapse after 6 months treated with anthracycline/taxane combination as first line therapy or first line anthracycline based therapy and second line taxane based therapy for advanced or metastatic disease
  * Adjuvant anthracycline based therapy followed by relapse within 6 months treated with first line taxane based therapy for advanced or metastatic disease
* Disease progression within 6 months of last taxane based chemotherapy
* No brain metastases
* Hormonal receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase and transaminases no greater than 2.5 times ULN (no greater than 5 times ULN in case of liver metastases)

Renal:

* Creatinine less than 1.25 times ULN

Cardiovascular:

* LVEF at least 50% if prior total dose of doxorubicin 550 mg/m2 or greater, epirubicin 900 mg/m2 or greater, or pirarubicin 700 mg/m2 or greater
* No prior or active congestive heart failure, myocardial infarction, or angina
* No uncontrolled hypertension or arrhythmia

Other:

* No unstable systemic disease
* No active infection
* No grade 2 or greater peripheral neuropathy
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior high dose chemotherapy with hematopoietic rescue
* No concurrent immunotherapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) for prevention of neutropenia

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 1 prior taxane based chemotherapy for advanced or metastatic disease
* No prior high dose chemotherapy with hematopoietic rescue
* No prior platinum based chemotherapy
* No prior taxane chemotherapy other than docetaxel or paclitaxel
* No prior adjuvant or neoadjuvant therapy with taxane/anthracycline based combination chemotherapy

Endocrine therapy:

* No concurrent steroids except in case of allergy prevention, emesis prophylaxis, or long term treatment for more than 3 months prior to study
* No concurrent hormonal anticancer therapy

Radiotherapy:

* No prior radiotherapy to study site unless evidence of disease progression
* Concurrent local radiotherapy allowed for pain relief

Surgery:

* At least 4 weeks since prior major surgery

Other:

* At least 4 weeks since prior anticancer and/or investigational drug
* No concurrent bisphosphonates unless started at least 2 months prior to study
* No other concurrent anticancer therapy
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-05; Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (10):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Institut Jules Bordet, Brussels (Bruxelles), Belgium
- France (3):
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Eugene Marquis, Rennes
- Universitats-Krankenhaus Eppendorf, Hamburg, Germany
- Israel (2):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom